CLINICAL TRIAL: NCT03047707
Title: Diagnostic Performance of S-Shearwave Elastography for Hepatic Fibrosis Evaluation: a Multicenter Prospective Study
Brief Title: S-Shearwave Elastography for Assessment of Hepatic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samsung Medison (Industry)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUH-2017-0215
Record Dates: First submitted 2017-02-08; First posted 2017-02-09 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Liver Fibroses
Keywords: ultrasound elastography; S-Shearwave; liver; fibrosis
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- S-Shearwave and TE (Experimental)
  Interventions: Diagnostic Test: S-Shearwave and TE

INTERVENTIONS:
Diagnostic Test: S-Shearwave and TE — S-Shearwave elastography and Transient elastography (TE) are performed to evaluate hepatic stiffness.

SUMMARY:
The purpose of this multi-center prospective study is to evaluate the diagnostic performance of S-Shearwave, a newly developed ultrasound shear wave elastography, for the assessment of hepatic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic liver disease or cirrhosis, or living-donor candidates for liver transplantation, or volunteers
* Signed informed consent

Exclusion Criteria:

* Acute hepatitis or bile duct obstruction
* Serum ALT> 5 times the upper limit of normal within 3 months
* s/p Rt. hemihepatectomy
* s/p liver transplantation
* Large mass or infiltrative lesion in the right lobe of the liver

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 634 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance to detect severe hepatic fibrosis (F3) | 3 months
  Reference standard: histologic diagnosis or Transient elastography

SECONDARY OUTCOMES:
Determination of cut-off values of S-Shearwave measurements for fibrosis grades according to causes | 3 months
Intra-observer and inter-observer agreement of S-Shearwave measurements | same day
Comparison of diagnostic performance: Shearwave vs. Transient elastography | 3 months
  Reference standard: histologic diagnosis
Usefulness of auto-profile function in S-Shearwave measurements | 3 months
Diagnostic value of B-mode ultrasound information for assessing hepatic fibrosis | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No